CLINICAL TRIAL: NCT04800562
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Efficacy and Safety of PCS499 in Treating Ulcerations in Patients Who Have Necrobiosis Lipoidica
Brief Title: A Clinical Trial to Evaluate PCS499 in Treating Ulcerations in Patients Who Have Necrobiosis Lipoidica
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of enrollment of this ultra rare disease
Sponsor: Processa Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PCS499-NL02
Record Dates: First submitted 2021-03-10; First posted 2021-03-16 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Necrobiosis Lipoidica
MeSH Terms: conditions — Necrobiosis Lipoidica

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PCS499 900mg BID (Experimental): PCS499 900mg twice a day with food
  Interventions: Drug: PCS499
- Placebo (Placebo Comparator): similar in appearance to active study drug
  Interventions: Other: placebo

INTERVENTIONS:
Drug: PCS499 — PCS499 900mg twice a day with food
  Arms: PCS499 900mg BID
Other: placebo — placebo comparator
  Arms: Placebo

SUMMARY:
This is a randomized, double blind, placebo controlled study that will evaluate the efficacy and safety of PCS499 as compared to placebo for the treatment of ulcerations of patients with necrobiosis lipoidica (NL) and will inform the design of future studies. Approximately 20 ulcerated NL patients who also meet other inclusion/exclusion criteria will be enrolled in the study. The primary objective of this study is to evaluate the efficacy of PCS499 as compared with placebo in ulcerated patients with Necrobiosis Lipoidica.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients age 18 to 80 years of age, inclusive, at Screening.
2. Biopsy-confirmed diagnosis of NL. Biopsies of continually active lesions performed outside of this clinical study will need to be reviewed and the diagnosis confirmed by the study pathologist. For patients with no previous history of biopsy, no biopsy within the previous 5 years, a biopsy that is not confirmed to be NL, or newly active lesion, a biopsy to confirm a diagnosis of NL will be performed at the Screening visit.
3. Ulcers on a single leg ("reference leg") at Baseline should consist of at least one (1) ulcer with a minimum ulcer surface area of 1 cm2, total ulcer area of a minimum of 2 cm2, and no more than 6 ulcers. If ulcers are present on both legs, the Investigator will select the "reference leg". The ulcer(s) on the reference leg ("reference ulcers") and all other ulcers associated with the patient's NL ("other ulcers") present at the Baseline visit will be followed in the study.
4. Women of childbearing potential must have a negative serum pregnancy test at the Screening Visit and a negative urine pregnancy test at Baseline before dosing. Women of childbearing potential must use one of the following acceptable methods of contraception throughout the study: oral contraceptive medication, intrauterine device (IUD), hormonal implants, injectable contraceptive medications, double-barrier methods, or tubal ligation.
5. Females who are postmenopausal (age-related amenorrhea >= 12 consecutive months and increased follicle-stimulating hormone [FSH] > 40 mIU/mL. If necessary to confirm postmenopausal status, an FSH will be drawn at Screening) or who have undergone hysterectomy or bilateral oophorectomy are exempt from pregnancy testing.
6. Male patients must be willing to use appropriate contraceptive measures and refrain from sexual activity with any female who is pregnant or lactating.
7. Patient must be willing and able to swallow whole tablets.
8. Patient must be willing and able to comply with study procedures.
9. Patient must be willing and able to provide signed, informed consent.

Exclusion Criteria:

1. Current or previous (within 4 weeks of Baseline) treatment with:

   1. Oral corticosteroids.
   2. Topical drugs (including prescription and over-the counter) on the reference leg. (Topical non-medicated moisturizer treatment products can be administered);
   3. Systemic pentoxifylline, theophylline, or cilostazol.
   4. Oral retinoid.
   5. Other systemic immunosuppressant or immunomodulatory drugs, including but not limited to calcineurin inhibitors (e.g., tacrolimus), thalidomide, apremilast, anti-malarials (e.g., hydroxychloroquine, chloroquine), cyclosporine, mycophenolate mofetil, azathioprine, methotrexate, etc.
2. Current or previous (within 12 weeks of Baseline) treatment with any biologic therapy (e.g., adalimumab, etanercept, infliximab, anakinra, etc.).
3. Phototherapy/photochemotherapy (NBUVB, UVB, PUVA) within 6 weeks prior to Baseline
4. Skin grafting, or other surgical procedure (other than debridement) within 6 weeks prior to Baseline.
5. History of drug allergy, including but not limited to pentoxifylline or other xanthine derivatives, or other allergy, which in the opinion of the Investigator, contraindicates participation.
6. Anticipated concurrent use of a strong CYP1A2 inhibiting drug, including but not limited to cimetidine and/or fluvoxamine, during the course of the study (after Screening).
7. Fever (>38°C), or chronic, persistent, or recurring infection(s) at Screening or Baseline.
8. Any infection requiring oral antimicrobial therapy within 2 weeks prior to Baseline or any infection requiring parenteral antibiotics or hospitalization within 12 weeks prior to Baseline. Any treatment for such infections must have been completed and the infection cured for at least 2 weeks prior to Baseline.
9. History of sarcoidosis, pyoderma gangrenosum, or any other disorder (in the judgment of the Investigator) that would interfere with the evaluation of NL or require protocol prohibited medication.
10. History of any life threatening infection or sepsis within 12 months of Baseline:
11. Clinically significant cardiac disease including but not limited to unstable angina, acute myocardial infarction within 6 months of Baseline, and arrhythmia requiring therapy.
12. Patient has QTc interval ≥ 480 milliseconds on Screening Electrocardiogram (ECG); a second Screening ECG may be done at investigator's discretion but the average of the two QTc screening intervals must not be ≥ 480 milliseconds.
13. History of cerebral hemorrhage, cerebrovascular accident, transient ischemic attack, gastrointestinal bleeding, or retinal hemorrhage within 6 months of Baseline.
14. Patient has active or history of neoplastic disease (except for adequately treated non-invasive basal cell and/or squamous cell carcinoma or carcinoma in situ of the cervix) within the past 5 years prior to Baseline.
15. Presence of clinically significant medical condition(s) including but not limited to: renal, hepatic, cardiovascular, hematological, gastrointestinal, endocrine, pulmonary, neurological, psychiatric, substance abuse, and/or any other clinically significant disease or disorder, which in the opinion of the Investigator (by its nature or by being inadequately controlled), may put the patient at risk due to participation in the study, influence the results of the study, and/or affect the patient's ability to complete the study.
16. History of or current diagnosis of active tuberculosis (TB); undergoing treatment for latent TB infection (LTBI); untreated LTBI (as determined by documented results within 3 months of the Screening Visit of a positive TB skin test with purified protein derivative with induration >= 5 millimeter (mm), or a positive QuantiFERON-TB test or positive or borderline T-Spot [Elispot] test); or positive TB test at Screening. Subjects with documented completion of appropriate LTBI treatment would not be excluded and are not required to be tested.
17. Vaccination with live or live-attenuated virus vaccine within 1 month prior to Baseline.
18. The results of the following laboratory tests performed at the central laboratory at Screening meet any of the criteria below:

    1. Hemoglobin < 8.0 g/dL (International System of Units (SI): < 80 g/L);
    2. White blood cells < 3.0 x 10^3 cells/mm^3 (SI: < 3.0 x 10^9 cells/L);
    3. Neutrophils < 1.0 x 10^3 cells/mm^3 (SI: < 1.0 x 10^9 cells/L);
    4. Lymphocytes < 0.5 x 10^3 cells/mm^3 (SI: < 0.5 x 10^9 cells/L);
    5. Platelets < 100 x 10^3 cells/mm^3 (SI: < 100 x 10^9 cells/L)
    6. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and/or alkaline phosphatase (ALP) ≥ 2 x upper limit of normal (ULN);
    7. Total bilirubin level ≥ 2 x ULN unless the individual has been diagnosed with Gilbert's disease and this is clearly documented;
    8. Estimated glomerular filtration rate < 40 mL/min/1.73 m^2 based on the Modification of Diet in Renal Disease (MDRD) formula.
    9. HbA1c > 10%
    10. Positive HIV serology
    11. Evidence of active Hepatitis B Virus (HBV) infection
    12. Evidence of active Hepatitis C Virus (HCV) infection
19. Women who are pregnant or breastfeeding.
20. Patient unwilling or unable to swallow tablets whole.
21. Any other medical condition, serious intercurrent illness, or extenuating circumstance that, in the opinion of the Investigator, would preclude participation in the study.
22. Use of any investigational product within 30 days prior to Baseline or currently enrolled in another study that involves clinical investigations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Incidence of ulcer closure as assessed by skin exam in patients treated with PCS499 as compared to placebo | ~ 6 months
  Evaluation of proportion of patients with wound closure based on skin evaluation in patients with NL as compared with placebo

CONTACTS AND LOCATIONS:
Overall Officials: Sian Bigora, PharmD, Study Director — Processa Pharmaceuticals
Locations (4):
- United States (4):
  - Processa Clinical Site, San Diego, California
  - Processa Clinical Site, Rochester, Minnesota
  - Processa Clinical Site, Charleston, South Carolina
  - Processa Clinical Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No